CLINICAL TRIAL: NCT03368014
Title: Community-based Mental Wellness Project for Adolescents and Adults: "Fun．Feel．Share" Lyrics-writing and Singing Show - A Pilot Project
Brief Title: "Fun．Feel．Share" Lyrics-writing and Singing Show
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Boys' and Girls' Clubs Association of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPH-MHP-BGCA02
Record Dates: First submitted 2017-09-04; First posted 2017-12-11 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Mental Health Wellness 1
Keywords: Sharing; Mind; Enjoyment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyrics-writing and singing show (Experimental): The one-hour lyrics-writing and singing workshop was conducted first at the beginning of the programme for the intervention group, followed by two small workshops teaching lyrics-writing skills and the lyrics-writing competition after the workshop. A lyrics writing and singing show and an award ceremony will be held at the end.
  Interventions: Behavioral: Lyrics-writing and singing show
- Waitlist control (No Intervention): The workshops will not be provided to the control schools during the evaluation period and will be provided after the evaluation period.

INTERVENTIONS:
Behavioral: Lyrics-writing and singing show — Participants will participate in a Lyrics-Writing and Singing Competition. They will first attend a lyrics-writing workshop and a short talk on SME (Sharing, Mind, Enjoyment) focusing on praising family members and knowledge of adolescent mental health problem (in particular the anxiety disorders) and mental well-being; submit SME (Sharing, Mind, Enjoyment) worksheet, such as "Express Your Love to Family Member" after the workshops; participate in the SME (Sharing, Mind, Enjoyment) Lyrics-writing and Singing Show and Award Ceremony (sharing) with a live performance by awarded entries and prize presentation ceremony.
  Arms: Lyrics-writing and singing show

SUMMARY:
"Fun．Feel．Share" Lyrics-writing and Singing Show - A Pilot Project is part of the Community-based Mental Wellness Project for Adolescents and Adults, which aims at promoting Sharing, Mind and Enjoyment (SME) and enhancing mental well-being. The Mental Wellness Project is financially supported by the Health Care and Promotion Fund from Food and Health Bureau and led by the School of Public Health, University of Hong Kong (HKU). "Fun．Feel．Share" Lyrics-writing and Singing Show - A Pilot Project aims to promote the SME related behaviors of adolescents through intervention of physical activities, and to promote their happiness, well-being and mental health knowledge.

DETAILED DESCRIPTION:
A cluster randomized controlled trial design will be adopted. The major subjects are 720-900 students. Four secondary schools in Hong Kong will be included in the evaluation. Schools will either be assigned into lyrics-writing and singing show intervention group or wait-list control group (the intervention won't be provided during the evaluation period and will be provided after the evaluation period).

The intervention mainly included 1) Lyrics-writing and Singing Competition with student and family entries: [a] lyrics-writing workshop and a short talk on SME focusing on praising family members and knowledge of adolescent mental health problem (in particular the anxiety disorders) and mental well-being; [b] use SME as theme for lyrics-writing and submit records of SME during lyrics-writing and singing; and [d] all entries are submitted in the form of audios. 2) SME Lyrics-writing and Singing Show and Award Ceremony (sharing): live performance by awarded entries and prize presentation ceremony.

There will then be 4 assessments (pre-intervention, immediate post intervention, one month and three months after baseline) to evaluate the effects of the intervention programme. In the assessments, students will be asked to complete questionnaires to measure the changes in SME related behaviors, happiness, well-being and knowledge and attitude towards mental health. The satisfaction towards the intervention, as well as the level of participation and ratings for the intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Students (major subjects): (Intervention group and waitlist control group)

  1. Chinese speaking
  2. Intact verbal and hearing abilities for interpersonal communication
  3. Reading and writing abilities for questionnaire completion
  4. Secondary school students
* Parents: (Intervention group)

  1. Chinese speaking
  2. Intact verbal and hearing abilities for interpersonal communication
  3. Reading and writing abilities for questionnaire completion
  4. With at least one secondary school child
* School principals/teachers/community partners: (Intervention group)

  1. Principals/teachers of intervention school and/or staffs of The Boys' and Girls' Clubs Association in partnership with HKU research team who organize plan or implement the project
  2. Adults aged 18 or above
  3. Chinese speaking
  4. Intact verbal and hearing abilities for interpersonal communication
  5. Reading and writing abilities for questionnaire/individual in-depth interviews completion

Exclusion Criteria:

* Students who cannot read Chinese

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1784 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in the concept of Sharing, Mind and Enjoyment (SME) for adolescents and their family members. | T1: before the lyrics-writing workshop (baseline); T3: after the lyrics-writing competition (2-month after baseline); T4: after the singing show and award ceremony (4-month after baseline)
  The outcome-based questionnaire will be used to evaluate participants' frequency of performing the suggested Sharing, Mind and Enjoyment (SME) related behaviors from baseline to four-month after baseline.

SECONDARY OUTCOMES:
Changes in the knowledge and understanding about mental health for adolescents and their family members. | T1: before the lyrics-writing workshop (baseline); T2: immediately after the workshop ( post intervention ); T3: after the lyrics-writing competition (2-month after baseline); T4: after the singing show and award ceremony (4-month after baseline)
  The outcome-based questionnaire will be used to evaluate participants' knowledge and understanding about anxiety disorder from baseline to four-month after baseline.
Changes in personal happiness from baseline to four-month after baseline | T1: before the lyrics-writing workshop (baseline); T3: after the lyrics-writing competition (2-month after baseline); T4: after the singing show and award ceremony (4-month after baseline)
  Personal Personal happiness will be assessed by Subjective Happiness Scale (SHS). SHS was rated on 7-point scale with 1 indicating not happiness at all and 7 indicating extreme happiness. To score the scale, the 4th item will be coded reversely and mean of the 4 items will be computed.
Changes in mental well-being from baseline to four-month after baseline. | T1: before the lyrics-writing workshop (baseline); T3: after the lyrics-writing competition (2-month after baseline); T4: after the singing show and award ceremony (4-month after baseline)
  Mental well-being will be assessed by validated Chinese version of 7-item Warwick Edinburgh Well-being Scale
Changes in individual and family health from baseline to four-month after baseline | T1: before the lyrics-writing workshop (baseline); T3: after the lyrics-writing competition (2-month after baseline); T4: after the singing show and award ceremony (4-month after baseline)
  Self-perceived health, happiness and harmony at the individual and family level will be assessed by a 0-10 score at 3 time points
Satisfaction toward "Fun．Feel．Share" Lyrics-writing and Singing Show Project | T2: immediately after the workshop ( post intervention ); T3: after the lyrics-writing competition (2-month after baseline); T4: after the singing show and award ceremony (4-month after baseline)
  Satisfaction towards the workshop, lyrics-writing competition, singing show and award ceremony will be assessed by programme evaluation measure
The social impact of the community-based engagement project | T4: after the singing show and award ceremony (4-month after baseline)
  The social impact of the community-based engagement project will be The satisfaction, ratings and opinions on "Fun．Feel．Share" Lyrics-writing and Singing Show programme of school principal/teacher/community partner in the intervention group will be assessed qualitatively (individual in-depth interviews)
The process of community based intervention programme | up to 4 months
  The process evaluation on-site observation questionnaire will be used to assess the process of the community-based intervention programs.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel, Sai Yin Ho, Dr., Principal Investigator — Associate Professor
Locations (1):
- School of Public Health, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03368014/Prot_SAP_000.pdf